CLINICAL TRIAL: NCT06652867
Title: Hypoglycemia Biomarkers to Predict Timing of a Hypoglycemic Event
Status: Completed | Type: Observational
Sponsor: Royal College of Surgeons in Ireland - Medical University of Bahrain (Other)
Collaborators: King Hamad University Hospital, Bahrain (Other)
Responsible Party: Sponsor
Other Study IDs: 400 / 05-Feb-2024
Record Dates: First submitted 2024-03-06; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Hypoglycemia
Keywords: type 1 Diabetes; Type 2 Diabetes; Hypoglycemia Biomarkers
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 5 ml of centrifuged serum blood sample will be retained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hypoglycemic diabetic patients: Hypoglycemic diabetic patients with type 1 or type 2 diabetes recruited during the incidence of hypoglycemia with awareness of the time when hypoglycemia occurred.
- Control group of non-hypoglycemic diabetic patients.: Type 1 or type 2 diabetic subjects who don't have hypoglycemia at the time of recruitment or in the last 72 hours.

SUMMARY:
The study aims to obtain a panel of biomarkers from hypoglycemic diabetic patients with either type 1 or type 2 diabetics and from control patients with type 1 or type 2 diabetes who didn't have hypoglycemia in the last 72 hours.

DETAILED DESCRIPTION:
Primary endpoint is establishing a panel of biomarkers from 100 hypoglycemic diabetic patients with type 1 or type 2 Diabetes during the incidence of hypoglycemia by taking a single blood sample to be analyzed for HbA1c, LDL, HDL, Triglycerides, CRP, CBC and biochemical analysis including liver and kidney function tests. In addition to 5 ml serum sample to be centrifuged and stored in RCSI lab.

Inpatient hypoglycemic patients may also be included in group of hypoglycemia and will be required to have a serial of blood samples taken to be analyzed on the 1st hour, 2nd hour, 3rd hour and 4th hour after the hypoglycemic event.

Secondary endpoint involves recruitment of 100 control Diabetic patients with type 1 or type 2 Diabetes to establish a panel of biomarkers by obtaining a blood sample for the HbA1c, LDL, HDL, Triglycerides, CRP, CBC and biochemical analysis including liver and kidney function tests to include 50 subjects fasting overnight and the other 50 subjects to be non-fasting but without having hypoglycemia at the time of recruitment or in the last 72 hours.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for diabetes subjects with hypoglycemia

* Diagnosed of type 2 diabetes or type 1 based on the WHO guidelines Patient's age from 21-75 years old
* Able to say when the hypo had occurred (free style libre in the outpatient setting, or documented blood glucose less than < 4 mmol/l (<70 mg/dl) as an inpatient

Inclusion criteria for diabetes subjects without hypoglycemia:

* Diagnosed of type 2 diabetes or type 1 based on the WHO guidelines
* Patient's age from 21-75 years old
* No hypoglycemia or hypoglycemia unawareness.

Exclusion Criteria:

* eGFR less than 45 ml/min
* Liver enzymes 3 folds greater than upper limit
* Pregnancy
* Patients on steroids or Atypical Antipsychotics or Cyclosporine/Tacrolimus or other medications that may mask hypoglycemia

Exclusion Criteria for diabetes subjects with hypoglycemia

* Unable to determine when hypoglycemic event had taken place
* Hypoglycemic unawareness
* Severe hypoglycemic event in the last 3 months

Exclusion criteria for diabetes subjects without hypoglycemia

* Hypoglycemic event in the preceding week
* Hypoglycemic unawareness

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type 1 or type 2 Diabetic subjects with and without hypoglycemic event to be included either in hypoglycemic group or in Control group.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-03-03 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Concentrations of a Panel of Protein Biomarkers in hypoglycemic subjects | 1 day from time of presentation
  a panel of biomarkers is measured from a blood test taken during the incidence of hypoglycemia from type 1 or type 2 Diabetic subject.

SECONDARY OUTCOMES:
Concentrations of a Panel of Protein Biomarkers Reference Ranges from non-hypoglycemic diabetic subjects | 3 days from time of presentation
  a panel of biomarkers is measured from a blood test taken from Diabetic subjects (type 1 or type 2) without having hypoglycemia.

OTHER OUTCOMES:
CBC | 1 day from time of presentation
  Measured from a blood test taken from Diabetic subjects (type 1 or type 2) control group and hypoglycemic patients
CRP | 1 day from time of presentation
  Measured from a blood test taken from Diabetic subjects (type 1 or type 2) control group and hypoglycemic patients
LDL | 1 day from time of presentation
  Measured from a blood test taken from Diabetic subjects (type 1 or type 2) control group and hypoglycemic patients
HDL | 1 day from time of presentation
  Measured from a blood test taken from Diabetic subjects (type 1 or type 2) control group and hypoglycemic patients
Triglycerides | 1 day from time of presentation
  Measured from a blood test taken from Diabetic subjects (type 1 or type 2) control group and hypoglycemic patients
Biochemical analysis | 1 day from time of presentation
  Measured from a blood test taken from Diabetic subjects (type 1 or type 2) control group and hypoglycemic patients
HbA1C% | 1 day from time of presentation
  Measured from a blood test taken from Diabetic subjects (type 1 or type 2) control group and hypoglycemic patients

CONTACTS AND LOCATIONS:
Overall Officials: Naji Alamuddin, Dr., Principal Investigator — Bahrain Royal Medical Services
Locations (1):
- Royal College of Surgeons in Ireland, Manama, Bahrain

IPD SHARING:
Plan to Share IPD: Yes
Monitoring, audits, and REC review will be permitted and provide direct access to source data and documents. The Lead PI and the researchers assigned by him will have access to the stored data/specimens. Only the Lead PI and the researchers assigned working on this study will be eligible to obtain the data/specimens from the participants during data collection
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Dr Naji will act as the data custodian and is responsible for the storage, handling and quality of the study data.
  Data will be collected in the case report form to allow for cross referencing to check validity.
  Study documents (paper and electronic) will be retained in a secure (kept locked when not in use) location during and after the trial has finished. All essential documents including source documents will be retained for a period of 3 years after study completion (last patient, last study point). A label stating the date after which the documents can be destroyed will be placed on the inside front cover of the case notes of trial participants.
Access Criteria: Study documents (paper and electronic) will be retained in a secure (kept locked when not in use) location during and after the trial has finished.

REFERENCES:
- [Background] Wei M, Gibbons LW, Mitchell TL, Kampert JB, Stern MP, Blair SN. Low fasting plasma glucose level as a predictor of cardiovascular disease and all-cause mortality. Circulation. 2000 May 2;101(17):2047-52. doi: 10.1161/01.cir.101.17.2047. PMID 10790345
- [Background] Goto A, Arah OA, Goto M, Terauchi Y, Noda M. Severe hypoglycaemia and cardiovascular disease: systematic review and meta-analysis with bias analysis. BMJ. 2013 Jul 29;347:f4533. doi: 10.1136/bmj.f4533. PMID 23900314
- [Background] Bonds DE, Miller ME, Bergenstal RM, Buse JB, Byington RP, Cutler JA, Dudl RJ, Ismail-Beigi F, Kimel AR, Hoogwerf B, Horowitz KR, Savage PJ, Seaquist ER, Simmons DL, Sivitz WI, Speril-Hillen JM, Sweeney ME. The association between symptomatic, severe hypoglycaemia and mortality in type 2 diabetes: retrospective epidemiological analysis of the ACCORD study. BMJ. 2010 Jan 8;340:b4909. doi: 10.1136/bmj.b4909. PMID 20061358
- [Background] Graveling AJ, Frier BM. Hypoglycaemia: an overview. Prim Care Diabetes. 2009 Aug;3(3):131-9. doi: 10.1016/j.pcd.2009.08.007. Epub 2009 Sep 24. PMID 19782016
- [Background] UK Hypoglycaemia Study Group. Risk of hypoglycaemia in types 1 and 2 diabetes: effects of treatment modalities and their duration. Diabetologia. 2007 Jun;50(6):1140-7. doi: 10.1007/s00125-007-0599-y. Epub 2007 Apr 6. PMID 17415551
- [Background] Henderson JN, Allen KV, Deary IJ, Frier BM. Hypoglycaemia in insulin-treated Type 2 diabetes: frequency, symptoms and impaired awareness. Diabet Med. 2003 Dec;20(12):1016-21. doi: 10.1046/j.1464-5491.2003.01072.x. PMID 14632703
- [Background] Chico A, Vidal-Rios P, Subira M, Novials A. The continuous glucose monitoring system is useful for detecting unrecognized hypoglycemias in patients with type 1 and type 2 diabetes but is not better than frequent capillary glucose measurements for improving metabolic control. Diabetes Care. 2003 Apr;26(4):1153-7. doi: 10.2337/diacare.26.4.1153. PMID 12663589
- [Background] Leiter LA, J.F. Y, Chiasson JL, Harris SB, Kleinstiver P, Sauriol L. Assessment of the impact of fear of hypoglycemic episodes on glycemic and hypoglycemia management. Canadian Journal of Diabetes. 2005;29:186-92.
- [Background] Brod M, Alolga SL, Meneghini L. Barriers to initiating insulin in type 2 diabetes patients: development of a new patient education tool to address myths, misconceptions and clinical realities. Patient. 2014;7(4):437-50. doi: 10.1007/s40271-014-0068-x. PMID 24958464
- [Background] Budnitz DS, Lovegrove MC, Shehab N, Richards CL. Emergency hospitalizations for adverse drug events in older Americans. N Engl J Med. 2011 Nov 24;365(21):2002-12. doi: 10.1056/NEJMsa1103053. PMID 22111719
- [Background] Peyrot M, Barnett AH, Meneghini LF, Schumm-Draeger PM. Insulin adherence behaviours and barriers in the multinational Global Attitudes of Patients and Physicians in Insulin Therapy study. Diabet Med. 2012 May;29(5):682-9. doi: 10.1111/j.1464-5491.2012.03605.x. PMID 22313123
- [Background] Kilpatrick ES, Rigby AS, Warren RE, Atkin SL. Implications of new European Union driving regulations on patients with Type 1 diabetes who participated in the Diabetes Control and Complications Trial. Diabet Med. 2013 May;30(5):616-9. doi: 10.1111/dme.12075. Epub 2013 Feb 28. PMID 23215789
- [Background] Hepburn DA, Frier BM. Hypoglycemia Unawareness in Patients with Insulin-Treated Diabetes-Mellitus. Saudi Medical Journal. 1991;12(3):182-90.
- [Background] Gold L, Ayers D, Bertino J, Bock C, Bock A, Brody EN, Carter J, Dalby AB, Eaton BE, Fitzwater T, Flather D, Forbes A, Foreman T, Fowler C, Gawande B, Goss M, Gunn M, Gupta S, Halladay D, Heil J, Heilig J, Hicke B, Husar G, Janjic N, Jarvis T, Jennings S, Katilius E, Keeney TR, Kim N, Koch TH, Kraemer S, Kroiss L, Le N, Levine D, Lindsey W, Lollo B, Mayfield W, Mehan M, Mehler R, Nelson SK, Nelson M, Nieuwlandt D, Nikrad M, Ochsner U, Ostroff RM, Otis M, Parker T, Pietrasiewicz S, Resnicow DI, Rohloff J, Sanders G, Sattin S, Schneider D, Singer B, Stanton M, Sterkel A, Stewart A, Stratford S, Vaught JD, Vrkljan M, Walker JJ, Watrobka M, Waugh S, Weiss A, Wilcox SK, Wolfson A, Wolk SK, Zhang C, Zichi D. Aptamer-based multiplexed proteomic technology for biomarker discovery. PLoS One. 2010 Dec 7;5(12):e15004. doi: 10.1371/journal.pone.0015004. PMID 21165148
- [Background] Suhre K, Arnold M, Bhagwat AM, Cotton RJ, Engelke R, Raffler J, Sarwath H, Thareja G, Wahl A, DeLisle RK, Gold L, Pezer M, Lauc G, El-Din Selim MA, Mook-Kanamori DO, Al-Dous EK, Mohamoud YA, Malek J, Strauch K, Grallert H, Peters A, Kastenmuller G, Gieger C, Graumann J. Connecting genetic risk to disease end points through the human blood plasma proteome. Nat Commun. 2017 Feb 27;8:14357. doi: 10.1038/ncomms14357. PMID 28240269
- [Background] Kraemer S, Vaught JD, Bock C, Gold L, Katilius E, Keeney TR, Kim N, Saccomano NA, Wilcox SK, Zichi D, Sanders GM. From SOMAmer-based biomarker discovery to diagnostic and clinical applications: a SOMAmer-based, streamlined multiplex proteomic assay. PLoS One. 2011;6(10):e26332. doi: 10.1371/journal.pone.0026332. Epub 2011 Oct 17. PMID 22022604